CLINICAL TRIAL: NCT04449432
Title: Goals for Reaching Optimal Wellness: GROWell
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Collaborators: Duke University (Other); Pattern Health (Unknown); National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 1399548; 1R01NR017659-01A1 (NIH)
Record Dates: First submitted 2020-06-23; First posted 2020-06-26 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-08

CONDITIONS: Pregnancy Related; Gestational Weight Gain; Postpartum Weight Retention; Overweight and Obesity
Keywords: pregnancy; gestational weight gain; postpartum weight retention; overweight; obesity; diet; mHealth; digital health
MeSH Terms: conditions — Gestational Weight Gain; Overweight; Obesity

STUDY DESIGN:
Intervention Model Description: Comparing intervention to active control
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GROWell (Interactive Obesity Treatment Approach) (Experimental): With Self-regulation Theory as the framework, the Interactive Obesity Treatment Approach Adapted for Pregnancy/Postpartum includes four components: (1) personalized goal setting, (2) daily support and educational messages, (3) self-monitoring of behavior with tailored feedback, and (4) skills training. Each component aligns with the self- regulatory processes shown in previous studies to be necessary for behavior change. All interactions with participants are via text using a cell phone.
  Interventions: Behavioral: GROWell (Interactive Obesity Treatment Approach)
- Attention Support Control (Active Comparator): The attention control will be delivered using text messaging to reduce the potential placebo effect that interacting with our mHealth system may have on pregnancy weight gain and postpartum weight loss. Information will be provided to control group participants that is specific to pregnancy, labor, delivery, and early infancy, but not to diet. Texts are specific to the participant's partner, pregnancy, employment, and breastfeeding plans/status.
  Interventions: Behavioral: Attention Support Control

INTERVENTIONS:
Behavioral: GROWell (Interactive Obesity Treatment Approach) — Personalized messaging via cell phone to support healthy eating behaviors during pregnancy and through 6 months postpartum
  Arms: GROWell (Interactive Obesity Treatment Approach)
Behavioral: Attention Support Control — Personalized messaging via cell phone to support healthy behaviors during pregnancy and through 6 months postpartum
  Arms: Attention Support Control

SUMMARY:
Despite the negative consequences to maternal-child health from women gaining too much weight during pregnancy, up to 62% of overweight and obese women gain more pregnancy weight than is recommended. This project will establish the efficacy of Goals for Reaching Optimal Wellness (GROWell), an mHealth tool for achieving appropriate pregnancy weight gain and promoting postpartum weight loss among women who enter pregnancy overweight or obese. GROWell will fill a gap in research and clinical care by providing a validated, standalone mHealth tool for weight control during pregnancy and postpartum, which is a currently lacking resource.

DETAILED DESCRIPTION:
Research attempts to prevent excess gestational weight gain, defined as gaining more weight during pregnancy than Institute of Medicine (IOM) guidelines for prepregnancy body mass index (BMI), have largely been unsuccessful. Roughly 62% of overweight and 45% of obese women still gain more weight than recommended, increasing risk for postpartum weight retention. Few mobile health (mHealth) interventions have been trialed to address pregnancy-associated weight gain, which is a missed opportunity. Adult women are high users of technology for general and pregnancy-specific health information seeking and sharing. To fill this gap, the long-term goal of this research is to disseminate into clinical practice a standalone mHealth tool that is effective for overweight and obese pregnant women to achieve gestational weight gain within IOM recommendations and return to prepregnancy weight after childbirth. The goal of this application is to test GROWell: Goals for Reaching Optimal Wellness, an innovative, mHealth tool based on Self-regulation Theory that investigators designed in pilot work to achieve appropriate gestational weight gain and safe postpartum weight loss. The investigators propose a blinded, randomized controlled trial to test the efficacy of GROWell compared to an attention control also developed in a pilot. Investigators will recruit 480 women ages 18-44 with prepregnancy BMI 25-<40 and 10-16 weeks gestation of a singleton, uncomplicated pregnancy. Block randomization based on BMI, race, and recruitment clinic will be used to assign participants equally to arm 1, GROWell (n=240), or arm 2, the attention control (n=240). Upon study enrollment and through 6 months postpartum, GROWell participants will receive daily text messages that provide tailored education, problem-solving skills, and support to aid their personalized dietary goals. Once weekly, participants self-monitor overall adherence to their goals using text messages that prompt them to report on how they did in the past week. When users respond to this prompt, they immediately receive a text with tailored feedback on their adherence and long-term progress toward their goals. Control participants will receive weekly texts that provide personalized self-care, pregnancy, labor, delivery, and early infancy education. The specific aims are to: (1) Compare the efficacy of GROWell to the attention control in reducing the proportion of women who gain excess gestational weight based on IOM guidelines (>25 lbs for overweight and >20 lbs for obese) controlling for demographics, parity, physical activity, diet quality, and depression/anxiety; and (2) Compare the efficacy of GROWell to the attention control in reducing postpartum weight retention at 6 months post-birth as measured by the proportion of women who are within 5% of their prepregnancy weight, controlling for demographics, parity, physical activity, diet quality, breastfeeding, and depression/anxiety. This research addresses PA 18-135 (Maternal Nutrition and Pre-pregnancy Obesity) and will provide an innovative, evidence-based, standalone mHealth tool to reduce excess gestational weight gain and postpartum weight retention among overweight and obese women, currently an unavailable resource.

ELIGIBILITY:
Inclusion Criteria:

* 10-16 weeks gestation of a confirmed pregnancy (i.e., ultrasound/heartbeat detected)
* Nulliparous or >12 months since previous birth
* Receive care at one of eight UC Davis Obstetric Clinics and plan to deliver at UC Davis Medical Center
* BMI >25 and <40 who are willing to receive and respond to texts using their own cell phone or a study-provided phone

Exclusion Criteria:

* Known pregnancy or fetal complications/high-risk status
* Multiple gestation
* Unable to read/write English
* BMI >40
* Current smokers
* Quit smoking <6 months prior to enrollment

Ages: 18 Years to 44 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 480 (Actual)
Dates: Start 2020-12-14 (Actual); Primary Completion 2024-01-26 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Gestational Weight Gain | Mid-study (25-30 weeks)
  Gestational weight gain will be calculated as: [weight(delivery) - weight(preconception)]. Women will be categorized as gaining excess gestational weight if they started pregnancy as overweight and gained more than 25 pounds or started pregnancy as obese and gained more than 20 pounds.
Postpartum Weight Retention | End of study (50-55 weeks)
  Postpartum weight retention will be calculated as: [weight(6 months postpartum) - weight(preconception)]. Women will be categorized as experiencing postpartum weight retention if postpartum weight at 6 months is greater than 1.05*preconception weight.

SECONDARY OUTCOMES:
Adherence to text-based self- monitoring | mid-study (25-30 weeks) and post-study (50-55 weeks)
  Measured cumulatively by week as the number of times a participant responds to weekly prompts to report on her progress to the number of times she was prompted, calculated to a percent separately for prenatal and postnatal periods.
Adherence to prescribed goals | mid-study (25-30 weeks) and post-study (50-55 weeks)
  Measured cumulatively by week as the proportion of goals for which a participant has "good adherence" during the previous week, defined as adhering to the goal 5/7 days, or >70%, calculated to a percent and separately for prenatal and postpartum periods.

OTHER OUTCOMES:
Delivery type | mid-study (25-30 weeks)
  Categorical as cesarean or vaginal delivery
Fetal growth abnormalities | mid-study (25-30 weeks)
  categorical as small-for-gestational age, large-for- gestational-age, macrosomia, or none.
Pregnancy complications | mid-study (25-30 weeks)
  categorical as gestational diabetes, hypertension, preeclampsia/eclampsia, placental abruption, fetal death, antepartum admission, preterm birth with and without NICU admission, none

CONTACTS AND LOCATIONS:
Overall Officials: Leigh Ann Simmons, PhD, Principal Investigator — University of California, Davis
Locations (1):
- UC Davis, Davis, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Simmons LA, Phipps JE, Whipps M, Smith P, Carbajal KA, Overstreet C, McLaughlin J, De Lombaert K, Noonan D. From hybrid to fully remote clinical trial amidst the COVID-19 pandemic: Strategies to promote recruitment, retention, and engagement in a randomized mHealth trial. Digit Health. 2022 Sep 25;8:20552076221129065. doi: 10.1177/20552076221129065. eCollection 2022 Jan-Dec. PMID 36185388
- [Derived] Simmons LA, Phipps JE, Overstreet C, Smith PM, Bechard E, Liu S, Walker C, Noonan D. Goals for Reaching Optimal Wellness (GROWell): A clinical trial protocol of a digital dietary intervention for pregnant and postpartum people with prenatal overweight or obesity. Contemp Clin Trials. 2022 Feb;113:106627. doi: 10.1016/j.cct.2021.106627. Epub 2021 Nov 20. PMID 34813963
- See also: Learn more or sign up for the study here! — https://studypages.com/s/healthy-pregnancy-study-720304/